CLINICAL TRIAL: NCT04252651
Title: Association of Cytokines With the Development of Complications in Burn and Toxic Epidermal Necrolysis (TENS) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Joseph M. Still Research Foundation, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: JMSRF-CYT-P04
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Inflammatory Response; Multi Organ Failure; Nosocomial Infection; Deep Vein Thrombosis
MeSH Terms: conditions — Multiple Organ Failure; Cross Infection; Venous Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood Draw: This study will involve blood draws to test for specific cytokines
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — This study will involve blood draws to test for specific cytokines

SUMMARY:
This study will involve blood draws to test for specific cytokines. The study goal is to gain a better understanding of the role of inflammatory response in the development of specific complications in burn and TENS patients.

ELIGIBILITY:
Inclusion Criteria:

* is ≥18 years of age
* has been admitted to the Joseph M. Still Burn Center at Doctors Hospital Augusta with a burn diagnosis, or TENS OR SJS diagnosis (confirmed or non-confirmed), with an expected length of stay to be at least 7 days
* the subject or their legally authorized representative is able to provide informed consent
* has a negative urine or serum pregnancy test at screening (if female and has potential for pregnancy)

Exclusion Criteria:

* is moribund, or in the opinion of the investigator is not expected to survive
* has sustained an electrical burn

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples size will be patients from the burn ICU.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cytokine Response that develops into complications | up to one year
  The number of burn and TENS patients that develop subsequent medical complications

CONTACTS AND LOCATIONS:
Overall Officials: Michael Quinn, MD, Principal Investigator — Joseph M. Still Research Foundation, Inc.
Locations (1):
- Joseph M. Still Burn Center at Doctors Hospital, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Study results will be analyzed, and study data presented at an appropriate related Congress meeting. Journal publication in a related peer-reviewed journal would be expected after presentation.